CLINICAL TRIAL: NCT06256042
Title: Effectiveness of Arthrocentesis and the Occlusal Splint in Treatment of Disc Displacements of the Temporomandibular Joint
Brief Title: Effectiveness of Arthrocentesis and the Occlusal Splint in Treatment of the TMJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Gustavo Grothe Machado, Director of Oral and Maxillofacial Surgery Service, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50207321.8.0000.0068
Record Dates: First submitted 2024-01-23; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Temporomandibular Joint Disc Displacement; Anterior Disc Displacement
Keywords: Temporomandibular joint; Anterior disc displacement; Arthrocentesis; Interocclusal stabilizing splint.
MeSH Terms: interventions — Occlusal Splints; Arthrocentesis

STUDY DESIGN:
Intervention Model Description: Stabilizing interocclusal plate (IOP): a stabilizing maxillary acrylic occlusal plate was made, flat, total and adjusted in central relation (RC). Advice and guidance on the disease.
  Arthrocentesis: Delimitation of a corner-tragus line to mark points A (10mm in front of the tragus and 2mm below the CT line) and B (20mm in front of the tragus and 10mm below the CT line); Local intra- and extra-oral antisepsis with aqueous chlorhexidine 0.12% and 0.2%, respectively; Local anesthesia of the auriculotemporal and intra-capsular nerve with mepivacaine 2% + Epinephrine 1:100,000; Insertion of the first 30x0.8 mm needle at point A and injection of 2-3 mL of Lactated Ringer; Insert the second 30x0.8 mm needle into point B Wash with 100-200mL of Ringer Lactate; Removal of the second needle; Injection of 1mL of 20mg Triamcinolone diluted in 0.9% saline solution (1:1) through the needle at point A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthrocentesis (Active Comparator): Delimitation of a corner-tragus line to mark points A (10mm in front of the tragus and 2mm below the CT line) and B (20mm in front of the tragus and 10mm below the CT line); Local intra- and extra-oral antisepsis with aqueous chlorhexidine 0.12% and 0.2%, respectively; Local anesthesia of the auriculotemporal and intra-capsular nerve with mepivacaine 2% + Epinephrine 1:100,000; Insertion of the first 30x0.8 mm needle at point A and injection of 2-3 mL of Lactated Ringer; Insert the second 30x0.8 mm needle into point B Wash with 100-200mL of Ringer Lactate; Removal of the second needle; Injection of 1mL of 20mg Triamcinolone diluted in 0.9% saline solution (1:1) through the needle at point A.
  Interventions: Procedure: Arthrocentesis
- Occlusal splint (Active Comparator): A stabilizing maxillary acrylic occlusal splint was made, flat, total and adjusted in central relation (RC).
  Interventions: Procedure: Occlusal splint

INTERVENTIONS:
Procedure: Occlusal splint — a stabilizing maxillary acrylic occlusal splint was made, flat, total and adjusted in central relation (RC).
  Arms: Occlusal splint
Procedure: Arthrocentesis — The patient then underwent arthrocentesis of the temporomandibular joint itself, following the Nitzan technique.
  Arms: Arthrocentesis

SUMMARY:
The goal of this clinical trial is to compare occlusal splint and arthrocentesis in patients with disc displacement with/without reduction. The main question it aims to answer are:

• Is there a more effective treatment for this cases?

Participants will answer a questionary about pain and functional limitations.

Researchers will compare Group 1(occlusal plate) and Gruoup 2 (arthrocentesis) to see if there is pain reduction and functional improvement in patients with disc displacement with/without reduction

DETAILED DESCRIPTION:
Introduction: Temporomandibular joint disc displacement is a disorder in which the articular disc is anteriorly displaced from its correct position in relation to the mandibular condyle and mandibular fossa. Traditionally, the initial treatment of disc displacements involves several conservative measures, among them, the stabilizing interocclusal splint. However, in cases where there is associated opening limitation, such as intermittent lock and closed-lock, arthrocentesis has been suggested as another initial treatment modality due to its faster effect in preventing disease progression to a more advanced stage, in addition to reducing the chances of pain chronicity and central sensitization. Objectives: The present study aimed to compare and analyze the effectiveness and benefits of performing arthrocentesis as the initial treatment in patients with DDWR with intermittent lock and in patients with DDWoR, compared to the stabilizing interocclusal splint. Additionally, it had as secondary objectives to characterize the sample according to demographic, systemic, local and psychosocial factors in both groups and to correlate the clinical characteristics of the included patients with the imaging findings of the MRI scans. Methods: A randomized, prospective, longitudinal pilot study was performed. The sample was obtained by convenience from a demand through consultations and referral, among patients treated at the Oral and Maxillofacial Surgery Service of HCFMUSP, from June 2021 to July 2023. Patients with diagnoses of: DDWR intermittent lock and DDWoR with opening mouth limitation. Study patients underwent an initial assessment using a clinical questionnaire (DC/TMD) and underwent an initial TMJ MRI. Then, they were randomly divided into two groups according to the treatment to which they would be submitted: stabilizing inter-occlusal splint (group 1) or arthrocentesis (group 2). After treatment was instituted, patients were evaluated at 1, 2, 3 and 6 months regarding clinical parameters of pain, functionality and psychosocial status.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old;
* Diagnosed with disc displacement with reduction with intermittent block or disc displacement without reduction;
* Availability of clinical follow-up for 6 months.

Exclusion Criteria:

* Pregnant patients;
* Patients undergoing conservative or invasive interventions to treat TMD in the last 6 months;
* Inability to use a stabilizing occlusal splint;
* Presence of toothache, neoplasms or medical contraindication for study participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Jaw function available in mouth opening and moviments of jaw | 6 months
  millimeter scale

SECONDARY OUTCOMES:
Pain available through of Visual Analogue Scale | 6 months
  the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10. It's been 0 (without pain) and 10 (worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo Faculty of Medicine Clinics Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No